CLINICAL TRIAL: NCT06182813
Title: The Effect of Binaural Auditory Beats on Hand-Eye Coordination in Adult Population.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FUI/CTR/2023/12
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Binaural Auditory Beats ,Hand-eye Coordination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- Experimental Group (Experimental): Group (A)/ Experimental group involves participants listening to the beta auditory beats for a duration of 25 min total.
  Out of these 25 minutes, the first 20 min will be spent while listening to the beta beats stimulus and the remaining 5 minutes will be used to carry out 3 trials of 30 seconds each with a rest period of 1 minute between each trial. The average values are taken for each participant out of the three trials. The number of successful catches are noted down for this test.
  Interventions: Other: Beta auditory beats (Group A)
- Group B- Control Group (Active Comparator): Group (B)/ Control group involves participants listening to the white noise for a duration of 25 min total.
  Out of these 25 minutes, the first 20 min will be spent while listening to the white noise stimulus and the remaining 5 minutes will be used to carry out 3 trials of 30 seconds each with a rest period of 1 minute between each trial. The average values are taken for each participant out of the three trials. The number of successful catches are noted down for this test.
  Interventions: Other: white noise (Group B)

INTERVENTIONS:
Other: Beta auditory beats (Group A) — Beta auditory beats for 25 min and then perform alternate wall toss test.
  Arms: Group A- Experimental Group
Other: white noise (Group B) — Involves participants receiving White noise for 25 min and then perform alternate wall toss test.
  Arms: Group B- Control Group

SUMMARY:
This research will deduce the effect of binaural auditory beats on Hand-Eye coordination and will further explore the connection between auditory binaural beats and potential health benefits whilst helping to raise awareness about the potential health benefits of binaural auditor beats among young adults.

The purpose of the study is to determine the effect of binaural auditory beats on hand-eye coordination in adult population.

This study will assess the effect of a beta acoustic beats with resultant frequency of 25 Hz and carrier frequencies of 385Hz in left ear and 410Hz β-acoustic frequency in corresponding right ear at the same time, The difference of magnitude of these two signals will provide the certain perceived wave frequency.

Each individual will be exposed to either beta auditory beats or white noise according to the group allotted.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To assess the effect of a beta acoustic beats with resultant frequency of 25 Hz and carrier frequencies of 385Hz in left ear and 410Hz β-acoustic frequency in corresponding right ear at the same time, the difference of magnitude of these two signals will provide the certain perceived wave frequency.
2. To compare the results of Hand-Eye Coordination for beta auditory beats and white noise.

HYPOTHESIS:

Alternate Hypothesis:

There is a significant effect of binaural auditory beats on hand-eye coordination in adult population. Null Hypothesis:

Null Hypothesis:

There is no significant effect of binaural auditory beats on hand-eye coordination in adult population.

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Rehabilitation department, Fauji Foundation Hospital Study duration: 18 months

Selection Criteria:

Inclusion Criteria Both genders (male and female) A healthy population with age limit 19-44yrs

Exclusion criteria:

Any person with blurred vision Any physical limitations or injuries that may hinder safe completion of activity.

If you have any reason to believe that you have difficulty processing sensory information.

Any other known condition or diagnoses that may affect cognition, attention, or hearing.

Regular cricket players

Sampling technique: Simple random sampling

Outcome Measures:

1. Data will be collected on Demographics and general information
2. The data will be collected through Audacity Software: for generating binaural acoustic beta beats and white noise. Alternate Wall Toss Test with validity and reliability of 0.718 and 0.875 respectively.

Experimental Group A = Before starting the actual trial participants will be informed about the protocols and the test procedure. The total duration of whole procedure is about 25 min. Out of these 25 minutes, the first 20 min will be spent while listening to the beta beats stimulus and the remaining 5 minutes will be used to carry out 3 trials of 30 seconds each with a rest period of 1 minute between each trial. The average values are taken for each participant out of the three trials. The number of successful catches are noted down for this test.

Control group (B) = The same procedure is taken out with white noise as a control group with the same tests and time duration.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study.

A printed questionnaire of inclusion criteria will be provided to the participants after obtaining written consent and providing adequate explanation regarding the study, after which the procedure is carried out.

Significance of the study:

This research will deduce the effects of binaural auditory beats on Hand-Eye coordination and will further explore the connection between auditory binaural beats and potential health benefits whilst helping to raise awareness about the potential health benefits of binaural auditor beats among young adults.

This study will add valuable evidence to the existing literature on binaural beat stimulation.

Most of the studies regarding beta beats focus on keeping your attention focused, analytical thinking and solving problems, stimulating energy and action, high-level cognition but there is a shortage of research focusing on the effects of beta auditory beats with coordination especially hand-eye coordination.

ELIGIBILITY:
Inclusion Criteria:

* Both genders (male and female)
* A healthy population with age limit 19-44yrs

Exclusion criteria:

* Any person with blurred vision
* Any physical limitations or injuries that may hinder safe completion of activity.
* If you have any reason to believe that you have difficulty processing sensory information.
* Any other known condition or diagnoses that may affect cognition, attention, or hearing.
* Regular cricket players

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Hand eye coordination using Alternate Wall toss test | Immediate after treatment(25 min)
  The scoring of Alternate wall toss test will be based on the score of the number of successful catches in a 30 second period.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan